CLINICAL TRIAL: NCT06126536
Title: Transcrestal Sinus Lift Using Osseodensification Versus Lateral Window Technique With Simultaneous Implant Placement
Brief Title: Transcrestal Sinus Lift Using Osseodensification Versus Lateral Window Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohammed Elsaid, Assistant Lecturer of Oral and Maxillofacial Surgery, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUAREC20190100-04
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Dental Implant; Sinus Lifting
Keywords: Osseodensification; Densah Burs; Internal Sinus lifting; External Sinus lifting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Crestal Maxillary Sinus Floor Elevation using Osseodensification: (Experimental): A crestal incision will be made towards the palate for better wound closure. A conservative flap will be raised, extending beyond the alveolar crest to minimize complications. In cases with 4-6mm ridge height and a need for 3mm vertical depth, a narrow densifying bur will be used, followed by wider burs to elevate the sinus membrane. The Densah® Bur will compact graft material to lift the membrane without penetrating the sinus floor. The osteotomy will be filled with bone graft substitute, and the final bur will apically propel the graft for vertical augmentation. Implant placement follows confirmation via radiography.
  Interventions: Procedure: Crestal Maxillary Sinus Floor Elevation using Osseodensification
- Group 2: Lateral Maxillary Sinus Floor Elevation (Experimental): In the Lateral technique, a crestal incision and mucoperiosteal flap will expose the sinus's lateral wall. A bony window is created, and when removable, sinus elevation curettes are used to elevate the sinus floor cautiously. Membrane perforations are covered with a resorbable collagen membrane if needed. Implant osteotomies follow standard protocol.
  Graft material mixed with saline is gently packed into the sinus to achieve the desired bone height. A resorbable membrane is placed on the window's outer surface, and the flap is sutured for primary closure.
  Interventions: Procedure: Lateral Maxillary Sinus Floor Elevation

INTERVENTIONS:
Procedure: Crestal Maxillary Sinus Floor Elevation using Osseodensification — Patients will be prepared for surgery with local anesthesia and thorough oral cavity disinfection. A full thickness crestal incision will be made slightly towards the palate to enhance the possibility of achieving primary wound closure. A conservative flap will be raised, extending slightly beyond the alveolar crest, to minimize flap-related issues. After preparing the osteotomy site using Densah burs and elevating the sinus to the desired height, the implant will be inserted into the osteotomy site.
  Arms: Group 1: Crestal Maxillary Sinus Floor Elevation using Osseodensification:
Procedure: Lateral Maxillary Sinus Floor Elevation — A crestal incision with an anterior vertical releasing incision exposes the sinus's lateral wall. A mucoperiosteal flap is carefully reflected, revealing the sinus. A bony window is created using a Piezoelectric device, and after elevation, the sinus floor is carefully lifted with various curettes. Implant osteotomies follow standard placement protocol, with precautions against sinus membrane perforation. Nanobone is used as graft material, mixed with saline and gently packed into the sinus. A resorbable membrane is placed on the window's outer surface, secured with circumferential resorbable sutures, and the flap is sutured for closure.
  Arms: Group 2: Lateral Maxillary Sinus Floor Elevation

SUMMARY:
The aim of this study is to evaluate the transcrestal sinus lift using Osseodensification versus lateral window technique with simultaneous implant placement.

DETAILED DESCRIPTION:
In Group 1, crestal maxillary sinus floor elevation will be done using Osseodensification. An incision will be made near the palate, and a conservative flap will be elevated. Osseodensification burs will be used to create an osteotomy and elevate the sinus membrane gradually. The osteotomy will be filled with bone graft, and the implant will be inserted.

In Group 2, lateral maxillary sinus floor elevation will be performed by creating a bony window in the lateral wall of the sinus. The sinus floor will be carefully elevated using sinus elevation curettes. If there's a membrane perforation, a collagen membrane will be applied. Bone substitute material will be packed into the sinus, and a resorbable membrane will be placed over the window before suturing.

Both groups will use Nanobone as the graft material.

ELIGIBILITY:
Inclusion Criteria:

* Patient with residual bone height from 4-6 mm and bone quality is D3 or D4.
* Patients had to require implant treatment in the posterior maxilla.
* All patients will sign a consent form before the study.

Exclusion Criteria:

* 1- Sinus pathology that precludes routine sinus augmentation.
* All contraindications of dental implants.11,12
* Heavy smokers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-12-07 (Actual); Primary Completion 2022-03-13 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Bone height gain | Immediate post-operative, 6 Months post-operative
  In Millimeter(mm)

SECONDARY OUTCOMES:
Ridge height | Immediate post-operative, 6 Months post-operative
  In Millimeter(mm)
Implant stability | Immediate post-operative, 6 Months post-operative
  In implant stability quotient (ISQ)
Bone Density | Immediate post-operative, 6 Months post-operative
  In Hounsfield units (HU)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine - Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Moraschini V, Uzeda MG, Sartoretto SC, Calasans-Maia MD. Maxillary sinus floor elevation with simultaneous implant placement without grafting materials: a systematic review and meta-analysis. Int J Oral Maxillofac Surg. 2017 May;46(5):636-647. doi: 10.1016/j.ijom.2017.01.021. Epub 2017 Feb 21. PMID 28254402
- [Background] Pjetursson BE, Tan WC, Zwahlen M, Lang NP. A systematic review of the success of sinus floor elevation and survival of implants inserted in combination with sinus floor elevation. J Clin Periodontol. 2008 Sep;35(8 Suppl):216-40. doi: 10.1111/j.1600-051X.2008.01272.x. PMID 18724852
- [Background] Jensen SS, Terheyden H. Bone augmentation procedures in localized defects in the alveolar ridge: clinical results with different bone grafts and bone-substitute materials. Int J Oral Maxillofac Implants. 2009;24 Suppl:218-36. PMID 19885447
- [Background] Chiapasco M, Casentini P, Zaniboni M. Bone augmentation procedures in implant dentistry. Int J Oral Maxillofac Implants. 2009;24 Suppl:237-59. PMID 19885448
- [Background] Summers RB. Sinus floor elevation with osteotomes. J Esthet Dent. 1998;10(3):164-71. doi: 10.1111/j.1708-8240.1998.tb00352.x. PMID 9759033
- [Background] Suk-Arj P, Wongchuensoontorn C, Taebunpakul P. Evaluation of bone formation following the osteotome sinus floor elevation technique without grafting using cone beam computed tomography: a preliminary study. Int J Implant Dent. 2019 Aug 1;5(1):27. doi: 10.1186/s40729-019-0181-7. PMID 31367919
- [Background] Kfir E, Goldstein M, Yerushalmi I, Rafaelov R, Mazor Z, Kfir V, Kaluski E. Minimally invasive antral membrane balloon elevation - results of a multicenter registry. Clin Implant Dent Relat Res. 2009 Oct;11 Suppl 1:e83-91. doi: 10.1111/j.1708-8208.2009.00213.x. Epub 2009 Aug 3. PMID 19681937
- [Background] Toffler M, Rosen P. Complications with transcrestal sinus floor elevation: Etiology, prevention, and treatment. In: Froum S (ed). Dental Implant Complications: Etiology, Prevention, and Treatment Hoboken, New Jersey: Wiley, 2015.
- [Background] Huwais S, Mazor Z, Ioannou AL, Gluckman H, Neiva R. A Multicenter Retrospective Clinical Study with Up-to-5-Year Follow-up Utilizing a Method that Enhances Bone Density and Allows for Transcrestal Sinus Augmentation Through Compaction Grafting. Int J Oral Maxillofac Implants. 2018 Nov/Dec;33(6):1305-1311. doi: 10.11607/jomi.6770. PMID 30427961
- [Background] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329